CLINICAL TRIAL: NCT03100903
Title: Safety, Tolerability, and Pharmacokinetics of Two Dose Strengths of a Single Subcutaneous Dose of BI 655130 and One Single Intravenous Dose of BI 655130 in Healthy Male and Female Subjects (Open-label, Parallel Group Design)
Brief Title: Safety, Tolerability, and Pharmacokinetics of a Subcutaneous and Intravenous Dose of BI 655130 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368.3; 2016-004557-32 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 655130 low dose SC (Experimental): Subject received single low dose BI 655130 solution as subcutaneous (SC) injection on day 1.
  Interventions: Drug: BI 655130
- BI 655130 high dose SC (Experimental): Subject received single high dose BI 655130 solution as subcutaneous (SC) injection on day 1.
  Interventions: Drug: BI 655130
- BI 655130 high dose IV (Experimental): Subject received single high dose BI 655130 solution as 30 minutes intravenous (IV) infusion on day 1.
  Interventions: Drug: BI 655130

INTERVENTIONS:
Drug: BI 655130 — single dose
  Other Names: Spesolimab

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of BI 655130 following subcutaneous administration (Test, T) compared to BI 655130 following intravenous infusion (Reference, R).

The secondary objective is the evaluation and comparison of several pharmacokinetic parameters between all tested treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP (Blood Pressure), PR (Pulse Rate)), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI (Body Mass Index) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and local legislation
* Male subjects, or female subjects who meet any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP (Blood Pressure), PR (Pulse Rate)), or ECG (Electrocardiogram),) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Female subjects will not be allowed to participate if any of the following applies:

* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Thoma C, Haeufel T, Li X. Assessment of the Pharmacokinetics and Safety of Spesolimab, a Humanised Anti-interleukin-36 Receptor Monoclonal Antibody, in Healthy Non-Japanese and Japanese Subjects: Results from Phase I Clinical Studies. Clin Pharmacokinet. 2022 Dec;61(12):1771-1787. doi: 10.1007/s40262-022-01176-5. Epub 2022 Dec 1. PMID 36451029
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, parallel group trial investigating two different dose strengths of a single subcutaneous (SC) dose of BI 655130 and one single intravenous (IV) dose of BI 655130.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Period: Overall Study
Arm/Group | BI 655130 Low Dose SC | BI 655130 High Dose SC | BI 655130 High Dose IV
Started | 12 | 12 | 12
Completed | 12 | 12 | 11
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS includes all subjects who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 655130 Low Dose SC | BI 655130 High Dose SC | BI 655130 High Dose IV | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (7.5) | 34.3 (8.1) | 38.6 (10.7) | 38.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 11 | 33
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 11 | 12 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 to the last quantifiable data point is presented. As defined in the statistical analysis plan, this outcome measure was analysed for comparison of subcutaneous (SC) versus intravenous (IV) administration of BI 655130 high dose as part of the primary analysis.
Time Frame: Pharmacokinetic samples were collected at pre-dose and at 0.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856, 3528 and 4200 hours after drug administration.
Population: Pharmacokinetic (PK) analysis set (PKS) restricted to high dose BI 655130 administration for primary analyses of the primary and secondary outcomes: All subjects of the Treated Set who were administered with BI 655130 high dose treatment and provided at least 1 observation for at least 1 primary or secondary PK endpoint that was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: Day*microgram/millilitre [day*μg/mL]
Arm/Group | BI 655130 High Dose SC | BI 655130 High Dose IV
Number analyzed (Participants) | 12 | 11
Day*microgram/millilitre [day*μg/mL] | 1579.19 (NA) — Adjusted geometric standard error = 1.07 | 2204.35 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: BI 655130 High Dose SC vs BI 655130 High Dose IV; Test type: Other — The statistical model was an analysis of variance (ANOVA) model on the logarithmic scale, accounting for the treatment group as a source of variation. The effect 'treatment group' was considered as fixed; Geometric Mean ratio (%) = 71.64, 90% CI 2-sided [60.57 to 84.73] — gMean ratio = gMean of BI 655130 high dose SC/gMean of BI 655130 high dose IV. Inter-individual geometric coefficient of variation (gCV) [%] = 23.7

2. Primary Outcome: Maximum Measured Concentration of BI 655130 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of BI 655130 in plasma is presented. As defined in the statistical analysis plan, this outcome measure was analysed for comparison of subcutaneous (SC) versus intravenous (IV) administration of BI 655130 high dose as part of the primary analysis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Microgram/millilitre [μg/mL]
Arm/Group | BI 655130 High Dose SC | BI 655130 High Dose IV
Number analyzed (Participants) | 12 | 11
Microgram/millilitre [μg/mL] | 33.36 (NA) — Adjusted geometric standard error = 1.08 | 113.90 (NA) — Adjusted geometric standard error = 1.08
Statistical Analysis 1: Comparison: BI 655130 High Dose SC vs BI 655130 High Dose IV; Test type: Other — [test comment as in outcome 1, analysis 1]; Geometric Mean (gMean) Ratio % = 29.29, 90% CI 2-sided [24.27 to 35.35] — gMean ratio = gMean of BI 655130 high dose SC/gMean of BI 655130 high dose IV. Inter-individual geometric coefficient of variation (gCV) [%] = 26.6

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 655130 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of BI 655130 in plasma over the time interval from 0 extrapolated to infinity is presented. As defined in the statistical analysis plan, this outcome measure was analysed for comparison of subcutaneous (SC) versus intravenous (IV) administration of BI 655130 high dose as part of the primary analysis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: Day*microgram/millilitre [day*μg/mL]
Arm/Group | BI 655130 High Dose SC | BI 655130 High Dose IV
Number analyzed (Participants) | 12 | 11
Day*microgram/millilitre [day*μg/mL] | 1600.92 (NA) — Adjusted geometric standard error = 1.07 | 2279.94 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: BI 655130 High Dose SC vs BI 655130 High Dose IV; Test type: Other — [test comment as in outcome 1, analysis 1]; Geometric Mean (gMean) Ratio % = 70.22, 90% CI 2-sided [59.26 to 83.20] — gMean ratio = gMean of BI 655130 high dose SC/gMean of BI 655130 high dose IV. Inter-individual geometric coefficient of variation (gCV) [%] = 23.9

ADVERSE EVENTS:
Time Frame: From first drug administration until end of the treatment, up to 179 days.
Description: Treated set (TS): TS includes all subjects who received study drug.
Arm/Group | BI 655130 Low Dose SC | BI 655130 High Dose SC | BI 655130 High Dose IV
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 11/12 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655130 Low Dose SC (N=12) | BI 655130 High Dose SC (N=12) | BI 655130 High Dose IV (N=12)
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 1
Sialoadenitis (Infections and infestations) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 3 | 1
Asthenia (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 1 | 0
Injection site induration (General disorders) | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03100903/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT03100903/SAP_001.pdf